CLINICAL TRIAL: NCT01103362
Title: Open-label Extension Trial for Pre- and Postmenopausal Women With HSDD
Brief Title: A 28-week Safety Study of Flibanserin in Pre- and Postmenopausal Women With Hypoactive Sexual Desire Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: administrative reasons
Sponsor: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 511.133
Record Dates: First submitted 2010-04-13; First posted 2010-04-14 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-04

CONDITIONS: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — flibanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- flibanserin 100mg (Experimental): flibanserin 100mg po qd
  Interventions: Drug: flibanserin

INTERVENTIONS:
Drug: flibanserin — all patients will receive open-label flibanserin 100mg

SUMMARY:
To generate additional long-term safety and efficacy data on flibanserin in premenopausal women and establish long-term safety and tolerability of flibanserin in naturally postmenopausal women with Hypoactive Sexual Desire Disorder who have completed a prior clinical trial of flibanserin (Trial 511.130, 511.147, or 511.156).

ELIGIBILITY:
Inclusion criteria:

1. Women with primary diagnosis of Hypoactive Sexual Desire Disorder (HSDD) who completed a prior trial of flibanserin. Such completion requires compliance with trial medication and the trial visit schedule including any post-treatment visits required in that clinical trial. Early discontinuation for any reason disqualifies the patient from entry into this trial. Patients must enroll in this study within 7 days after completing the final visit of the parent trial.
2. The premenopausal patient must use a medically acceptable method of contraception for at least two months before baseline and continue to use medically acceptable method of contraception during the trial.
3. Postmenopausal patients must be a naturally postmenopausal woman of any age with at least one ovary. Natural menopause is defined as greater than 12 months of spontaneous amenorrhea.
4. In the investigator's opinion, patients must be willing to adhere to trial requirements as well as to be able to perform them.
5. Patients must be able and willing to give meaningful, written informed consent prior to participation in the trial, in accordance with regulatory requirements. Patients must have sufficient understanding to communicate effectively with the investigator, and be willing to discuss sexual functioning with study staff.

Exclusion criteria:

1. Patients with history of Major Depressive Disorder (MDD) within six months prior to the Screen Visit, or a score of greater than or equal to 14 on the Beck Depression Inventory II (BDI-II), or a history of suicidal behavior or suicidal ideation according to the Columbia-Suicide Severity Rating Scale (C-SSRS®). If a psychiatrist or psychologist, using clinical judgment, believes a patient who scored between 14 and 19 on the BDI®-II is not depressed, the patient may be entered into the trial. NOTE: If a patient reports positive response to BDI®-II Question 9 and/or a Yes response to either C-SSRS® Suicide Ideation section Question 1 and/or 2 and/or any question in the Suicide Behavior section, please refer to Section 5.2.5 for immediate actions required.
2. At the Screen Visit, serum alanine aminotransferase, serum aspartate aminotransferase, alkaline phosphatase, or total bilirubin greater than or equal to three times upper limit of normal; blood urea nitrogen greater than or equal to 30 mg/deciliter (dL), plasma creatinine greater than or equal to 2 mg/dL, hemoglobin <9.5 grams/dL, leukopenia (<2.5 x 103/microliter [µL]), neutropenia (<1.5 x 103/µL), lymphopenia (<0.8 x 103/µL), thrombocytopenia (<100 x 103/µL) or thrombocytosis (>500 x 103/µL); or random glucose > upper limit of normal.
3. Patients with newly developed, self-reported symptoms after the End of Treatment parent trial visit and at this trial Screen Visit of pelvic inflammatory disease, urinary tract or vaginal infection / vaginitis, cervicitis, interstitial cystitis, vulvodynia, or significant vaginal atrophy.
4. Patients with history of any cancer within the last ten years, other than non-invasive, previously resected basal cell carcinoma of the skin.
5. Patients whose sexual function was affected by hysterectomy, oophorectomy, or any other pelvic or vaginal surgery.
6. Patients who are pregnant (by urine pregnancy test at the Screen Visit) or have been pregnant within the month prior to the Screen Visit or who are breast-feeding or have breast-fed within the last six months prior to the Baseline Visit.
7. Patients receiving medication excluded in their prior safety and efficacy trial of flibanserin causing sexual dysfunction or safety-relevant interactions (i.e., antidepressants, anxiolytics, antipsychotics, anticonvulsants, anticoagulants).
8. Patients with clinically relevant conditions which might interfere with their ability to participate in the trial.
9. Participation in a trial of an investigational medication other than flibanserin within one month prior to the Screen Visit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sprout Pharmaceuticals, Study Chair — Sprout Pharmaceuticals
Locations (95):
- United States (88):
  - 511.133.01074 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 511.133.01141 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 511.133.01046 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 511.133.01042 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 511.133.01025 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 511.133.01073 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 511.133.01127 Boehringer Ingelheim Investigational Site, Tuscon, Arizona
  - 511.133.01030 Boehringer Ingelheim Investigational Site, Encinitas, California
  - 511.133.01028 Boehringer Ingelheim Investigational Site, Fair Oaks, California
  - 511.133.01037 Boehringer Ingelheim Investigational Site, Irvine, California
  - 511.133.01136 Boehringer Ingelheim Investigational Site, La Mesa, California
  - 511.133.01128 Boehringer Ingelheim Investigational Site, Newport Beach, California
  - 511.133.01115 Boehringer Ingelheim Investigational Site, Oceanside, California
  - 511.133.01022 Boehringer Ingelheim Investigational Site, Sacremento, California
  - 511.133.01035 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.133.01052 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.133.01099 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.133.01016 Boehringer Ingelheim Investigational Site, Tarzana, California
  - 511.133.01021 Boehringer Ingelheim Investigational Site, Vista, California
  - 511.133.01051 Boehringer Ingelheim Investigational Site, Westlake Village, California
  - 511.133.01071 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 511.133.01053 Boehringer Ingelheim Investigational Site, Farmington, Connecticut
  - 511.133.01015 Boehringer Ingelheim Investigational Site, Groton, Connecticut
  - 511.133.01139 Boehringer Ingelheim Investigational Site, New London, Connecticut
  - 511.133.01064 Boehringer Ingelheim Investigational Site, Newark, Delaware
  - 511.133.01062 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 511.133.01003 Boehringer Ingelheim Investigational Site, Boynton Beach, Florida
  - 511.133.01056 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 511.133.01132 Boehringer Ingelheim Investigational Site, Coral Gables, Florida
  - 511.133.01065 Boehringer Ingelheim Investigational Site, Daytona Beach, Florida
  - 511.133.01020 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 511.133.01024 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 511.133.01043 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 511.133.01070 Boehringer Ingelheim Investigational Site, Palm Harbor, Florida
  - 511.133.01019 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 511.133.01061 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 511.133.01066 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 511.133.01001 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 511.133.01002 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 511.133.01009 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 511.133.01023 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 511.133.01082 Boehringer Ingelheim Investigational Site, Marietta, Georgia
  - 511.133.01008 Boehringer Ingelheim Investigational Site, Sandy Springs, Georgia
  - 511.133.01044 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 511.133.01034 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 511.133.01100 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 511.133.01067 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 511.133.01013 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 511.133.01031 Boehringer Ingelheim Investigational Site, Bingham Farms, Michigan
  - 511.133.01006 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 511.133.01014 Boehringer Ingelheim Investigational Site, Billings, Montana
  - 511.133.01060 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 511.133.01057 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 511.133.01039 Boehringer Ingelheim Investigational Site, Moorestown, New Jersey
  - 511.133.01017 Boehringer Ingelheim Investigational Site, Endwell, New York
  - 511.133.01135 Boehringer Ingelheim Investigational Site, Cary, North Carolina
  - 511.133.01047 Boehringer Ingelheim Investigational Site, New Bern, North Carolina
  - 511.133.01027 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 511.133.01138 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 511.133.01119 Boehringer Ingelheim Investigational Site, Fargo, North Dakota
  - 511.133.01033 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.133.01004 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 511.133.01050 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 511.133.01059 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 511.133.01058 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 511.133.01105 Boehringer Ingelheim Investigational Site, Englewood, Ohio
  - 511.133.01072 Boehringer Ingelheim Investigational Site, Edmond, Oklahoma
  - 511.133.01007 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 511.133.01055 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 511.133.01068 Boehringer Ingelheim Investigational Site, Mt. Pleasant, South Carolina
  - 511.133.01084 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 511.133.01063 Boehringer Ingelheim Investigational Site, Knoxville, Tennessee
  - 511.133.01010 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 511.133.01036 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 511.133.01018 Boehringer Ingelheim Investigational Site, Corpus Christi, Texas
  - 511.133.01032 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 511.133.01011 Boehringer Ingelheim Investigational Site, Katy, Texas
  - 511.133.01012 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.133.01026 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.133.01005 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 511.133.01069 Boehringer Ingelheim Investigational Site, Sandy City, Utah
  - 511.133.01040 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 511.133.01029 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.133.01075 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.133.01049 Boehringer Ingelheim Investigational Site, Virgnia Beach, Virginia
  - 511.133.01054 Boehringer Ingelheim Investigational Site, Renton, Washington
  - 511.133.01045 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 511.133.01038 Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Canada (7):
  - 511.133.02004 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 511.133.02014 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 511.133.02006 Boehringer Ingelheim Investigational Site, Burlington, Ontario
  - 511.133.02005 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 511.133.02016 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 511.133.02002 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 511.133.02003 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Simon JA, Derogatis L, Portman D, Brown L, Yuan J, Kissling R. Flibanserin for Hypoactive Sexual Desire Disorder: An Open-Label Safety Study. J Sex Med. 2018 Mar;15(3):387-395. doi: 10.1016/j.jsxm.2017.12.016. PMID 29502984

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flibanserin 100mg
Started | 596
Completed | 0
Not Completed | 596
Not completed — study terminated | 596

BASELINE CHARACTERISTICS:
Arm/Group | Flibanserin 100mg
Number analyzed (Participants) | 596
Age, Customized [Mean (Standard Deviation); unit: years]
  age | 45.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 596
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 473
  White Hispanic | 53
  Black/African American | 53
  Black/African American Hispanic | 1
  Asian | 7
  American Indian/Alaskan Native | 7
  Hawaiian/Pacific Islander | 2

OUTCOME MEASURES:

1. Primary Outcome: The Frequency of Adverse Events
Time Frame: A 28-week, open-label, safety, extension trial of flibanserin in premenopausal and postmenopausal women with HSDD
Measure: Number; unit: percentage of patients-any adverse event
Arm/Group | Flibanserin 100mg
Number analyzed (Participants) | 596
percentage of patients-any adverse event | 59.2

ADVERSE EVENTS:
Arm/Group | Flibanserin 100mg
Serious Adverse Events (participants affected / at risk) | 4/596
Other Adverse Events (participants affected / at risk) | 170/596
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 100mg (N=596)
Cellulitis (Infections and infestations) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin 100mg (N=596)
Dizziness (Nervous system disorders) | 57 (63)
somnolence (Nervous system disorders) | 47 (49)
Insomnia (Psychiatric disorders) | 34 (34)
Nausea (Gastrointestinal disorders) | 32 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No